CLINICAL TRIAL: NCT06063265
Title: Effect of a Six-week Integrated Attention Training Program on the Cognitive Functions of Older Adults With Co-occurring Anxiety Symptoms and Subjective Cognitive Complaints
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HMRF 10211426
Record Dates: First submitted 2023-08-29; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-08

CONDITIONS: Anxiety
Keywords: Subjective cognitive complaints; Attention training
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IATP (Experimental)
  Interventions: Behavioral: Integrated Attention Training Program
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Integrated Attention Training Program — Integrated Attention Training Program (IATP) specifically aims at training attentional control, which involves the coordination of complex behaviours, such as planning, reasoning, selection and information inhibition.
  Arms: IATP

SUMMARY:
The goal of this single-blind randomized control trial is to compare a 6-week Integrated Attention Training Program (IATP) and health education in older people with co-occurrence of anxiety symptoms and subjective cognitive decline (SCC).

The study aims to answer if a 6-week Integrated Attention Training Program (IATP) will improve cognitive, anxiety, and level of pro-inflammatory biomarkers in this high-risk group.

Older adults with co-occurring anxiety and SCC will be recruited to participate in a 6-week single-blind randomized controlled trial. IATP group (Intervention group) will undergo attention and functional training. Control group will receive health education.

Investigators will compare the IATP with health education to see if cognitive function, anxiety symptoms, and level of pro-inflammatory biomarkers in comparison to health education will improved after intervention and over 24 weeks.

DETAILED DESCRIPTION:
This is a 2-armed randomized control trial. For both groups, participants will attend a 45-minute training twice a week for consecutive 6 weeks in a group of 6 people. IATP group (I) will begin with 5 minutes of warm up to give instructions, followed by 5 minutes of breathing exercises, 5 minutes of body scanning, 10 minutes of dual-task training, 15 minutes of functional training, and 5 minutes of performance appraisal under guidance of an intervention instructor. Control group (C) will receive 12 sessions of health education on managing chronic diseases or conditions commonly found in old age during the intervention period.

Assessments will take place at baseline (T0), immediately after intervention (T1) and after 24-week (T2).

Measurement will include a battery of cognitive assessments, Hamilton Anxiety Scale (HAM-A), and a questionnaire on sociodemographic characteristics (age, sex, educational level, and socioeconomic status), physical and mental health statuses, and lifestyle patterns (smoking, drinking, and leisure activities in the past one month). In addition, a 15ml blood sample will be collected from each consenting participant by a phlebotomist for an inflammatory assay analysis at T0. Follow-up assessments and blood collections will be arranged at 6th (T1) and 24th (T2) week.

Linear mixed effects models will analyze the changes on anxiety and cognitive performance from baseline to endpoints. All the analyses will be based on Intention-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

1. Older adults aged 60 to 90 years;
2. No Major Neurocognitive Disorders
3. Presence of anxiety symptoms
4. Presence of Subjective Cognitive Complaints

Exclusion Criteria:

1. Clinical dementia
2. History of major depression
3. Presence of major neurological deficit
4. Presence of severe visual impairment; or
5. Currently on any psychotropic or other medications known to affect cognition; or
6. Participation in other cognitive trainings or interventions 6 months prior to this study or during the study period.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Attention - Digit Span Forward Task | 6 weeks after baseline and 6 months after baseline
  Participants are asked to repeat a series of digits immediately after presentation, in ascending order starting from 3 and up to 8 digits. Analysis of scoring is based on the span length achieved.
Attention - Chinese Trail Making Test - Part A (CTMT-A) | 6 weeks after baseline and 6 months after baseline
  The participant will need to connect between Arabic and Chinese numbers in sequential order. The completion time (in second) and the numbers of errors made during the test are recorded
Executive function - Category Verbal Fluency Test (CVFT) | 6 weeks after baseline and 6 months after baseline
  It is test of semantic fluency and executive function. Participants were asked to generate as many exemplars as possible for each of the three semantic categories, namely animals, fruits, and vegetables, in 60 seconds. Their responses were recorded in serial order. Analysis of scoring is based on the total number of words that the participant is able to produce across all three categories.
Executive function - Digit Span Backwards Task | 6 weeks after baseline and 6 months after baseline
  Participants will be asked to repeat a series of digits immediately after presentation, in reverse order starting from 2 and up to 8 digits. Analysis of scoring is based on the span length achieved.
Executive function - Chinese Trail Making Test - Part B (CTMT-B) | 6 weeks after baseline and 6 months after baseline
  The participant will need to connect and alternate between Arabic and Chinese numbers. The completion time (in second) and the numbers of errors made during the test are recorded.
Anxiety symptoms | 6 weeks after baseline and 6 months after baseline
  Hamilton Anxiety Scale (HAM-A) - each item will be scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where 17 or less indicates a mild severity, 18-24 indicates a mild to moderate severity and 25-30 a moderate to severe severity.
Level of inflammation | 6 weeks after baseline and 6 months after baseline
  Levels of IL-1β
Level of inflammation | 6 weeks after baseline and 6 months after baseline
  Levels of IL-6
Level of inflammation | 6 weeks after baseline and 6 months after baseline
  Levels of TNF-α
Level of inflammation | 6 weeks after baseline and 6 months after baseline
  Levels of CRP

SECONDARY OUTCOMES:
Functional performance - Chinese version of Disability of Assessment in dementia (CDAD) | 6 weeks after baseline and 6 months after baseline
  It is subdivided into basic activities of daily living (BADL) and instrumental activities of daily living (IADL). It evaluates the ability of an individual to initiate, plan and execute everyday activities. The overall score of DAD ranges from 0 to 100, with higher score indicating better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Ada WT FUNG, PhD, Principal Investigator — Hong Kong Baptist University
Locations (1):
- Ada WT FUNG, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No
Dissimination through conference presentation and publications